CLINICAL TRIAL: NCT05673356
Title: Anterior Cruciate Ligament Reconstruction With Quadriceps Tendon Bone Autograft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Artromedical Konrad Malinowski Clinic (Other)
Responsible Party: Principal Investigator, Konrad Malinowski MD, Konrad Malinowski MD, Artromedical Konrad Malinowski Clinic, Artromedical Konrad Malinowski Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-pro-ar-2022
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Anterior Cruciate Ligament Tear; Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Single Group: Clinical trials with a single arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm of the study (Experimental): Arthroscopic anterior cruciate ligament reconstruction with quadriceps tendon bone autograft (QTB) will be performed in these patients.
  Interventions: Procedure: Arthroscopic anterior cruciate ligament reconstruction with quadriceps tendon bone autograft (QTB)

INTERVENTIONS:
Procedure: Arthroscopic anterior cruciate ligament reconstruction with quadriceps tendon bone autograft (QTB) — Arthroscopic anterior cruciate ligament reconstruction with quadriceps tendon bone autograft (QTB) will be performed in these patients. QTB autografts will be harvested as described in the published technique: K. Malinowski, J. Paszkowski, M. Mostowy, A. Góralczyk, R.F. LaPrade, K. Hermanowicz, Quadriceps Tendon-Bone Full-Thickness Autograft: Reproducible and Easy Harvesting Technique Using Simple Surgical Tools, Arthrosc. Tech. 10 (2021) e1165-e1172. https://doi.org/10.1016/j.eats.2021.01.003. ACLR will be performed utilizing anteromedial technique with management of any accompanying intraarticular lesions.

SUMMARY:
Anterior cruciate ligament injuries are one of the most common sports knee injuries. Their effect on the knee joint can be detrimental with patients experiencing instability and progressive damage of the intraarticular structures. Therefore, anterior cruciate ligament reconstruction (ACLR) is often indicated. Multiple graft option exist, including autograft, allograft and xenograft tissues, with autografts being considered as a first-choice source of reconstructed ligament in most cases. Two most common harvested autografts are hamstring tendons (semitendinosus or semitendinosus and gracilis tendons; ST or STG) and patellar tendon with two bone blocks (bone - patellar tendon - bone; BPTB). However, in the recent literature there is an increasing trend towards use of quadriceps tendon autograft (QT). Multiple techniques of harvesting this graft were described, including both partial and complete thickness of the tendon. Another issue is whether bone block from the upper pole of the patella is harvested along with the soft tissues (quadriceps tendon bone graft, QTB).

The aim of this study is to add to the body of knowledge concerning full-thickness quadriceps tendon-bone autograft (QTB) used in ACLR. The primary outcome consists of The International Knee Documentation Committee Questionnaire (IKDC), the Knee injury and Osteoarthritis Outcome Score (KOOS) and retear rate.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee anterior and rotatory instability after ACL injury;
* Primary ACLR cases

Exclusion Criteria:

* Active inflammation of the knee;
* Revision cases;
* Additional PLC, PCL or PFJ injuries (MCL and meniscal lesions are not exclusion criteria);
* Fractures around the knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee stability | At the 12 month of the follow-up.
  Anterior and anterolateral rotatory knee stability assessed by the means of instrumented Lachman test and pivot-shift test.
Knee stability | At the 24 month of the follow-up.
  Anterior and anterolateral rotatory knee stability assessed by the means of instrumented Lachman test and pivot-shift test.

SECONDARY OUTCOMES:
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 12 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 24 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 12 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 24 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
Retear rate | At the 12 month of the follow-up.
  Rate of patients with retear of the reconstructed ligament
Retear rate | At the 24 month of the follow-up.
  Rate of patients with retear of the reconstructed ligament
ROM | At the 12 month of the follow-up.
  Knee range of motion assessed by the means of goniometer.
ROM | At the 24 month of the follow-up.
  Knee range of motion assessed by the means of goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Malinowski, MD PhD, Principal Investigator — Artromedical Orthopaedic Clinic, Bełchatów, Poland
Locations (1):
- Artromedical Orthopaedic Clinic, Bełchatów, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malinowski K, Paszkowski J, Mostowy M, Goralczyk A, LaPrade RF, Hermanowicz K. Quadriceps Tendon-Bone Full-Thickness Autograft: Reproducible and Easy Harvesting Technique Using Simple Surgical Tools. Arthrosc Tech. 2021 Mar 18;10(4):e1165-e1172. doi: 10.1016/j.eats.2021.01.003. eCollection 2021 Apr. PMID 33981566
- [Background] Lind M, Nielsen TG, Soerensen OG, Mygind-Klavsen B, Fauno P. Quadriceps tendon grafts does not cause patients to have inferior subjective outcome after anterior cruciate ligament (ACL) reconstruction than do hamstring grafts: a 2-year prospective randomised controlled trial. Br J Sports Med. 2020 Feb;54(3):183-187. doi: 10.1136/bjsports-2019-101000. Epub 2019 Nov 8. PMID 31704697
- [Background] Slone HS, Romine SE, Premkumar A, Xerogeanes JW. Quadriceps tendon autograft for anterior cruciate ligament reconstruction: a comprehensive review of current literature and systematic review of clinical results. Arthroscopy. 2015 Mar;31(3):541-54. doi: 10.1016/j.arthro.2014.11.010. Epub 2014 Dec 25. PMID 25543249
- [Background] Mehran N, Damodar D, Shu Yang J. Quadriceps Tendon Autograft in Anterior Cruciate Ligament Reconstruction. J Am Acad Orthop Surg. 2020 Jan 15;28(2):45-52. doi: 10.5435/JAAOS-D-19-00032. PMID 31305357
- [Background] Lund B, Nielsen T, Fauno P, Christiansen SE, Lind M. Is quadriceps tendon a better graft choice than patellar tendon? a prospective randomized study. Arthroscopy. 2014 May;30(5):593-8. doi: 10.1016/j.arthro.2014.01.012. Epub 2014 Mar 14. PMID 24630956